CLINICAL TRIAL: NCT02984995
Title: Phase 2 Open-label, Single-arm Study of Quizartinib (AC220) Monotherapy in Japanese Patients With FLT3-ITD Positive Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Phase 2 Study of Quizartinib in Participants With Acute Myeloid Leukemia (AML) FLT3 Internal Tandem Duplication (FLT3/ITD) Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-J201; JAPIC CTI-163441 (Other: JAPIC CTI)
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: FLT3-ITD; Positive refractory or relapsed acute myeloid leukemia; Hematology malignancy; Developmental Phase II
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Initial dose 30 mg/day quizartinib (Experimental): Participants who received an initial dose of 30 mg/day of quizartinib and, if no QT prolongation, the dose escalated to 60 mg/day at Day 15.
  Interventions: Drug: Quizartinib
- Initial dose 20 mg/day quizartinib (Experimental): Participants who received a CYP3A4 strong inhibitor received an initial dose of 20 mg/day of quizartinib and, if no QT prolongation, the dose escalated to 30 mg/day at Day 15.
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Quizartinib — Quizartinib was orally administered once daily every morning. Treatment with quizartinib was administered in 28-day cycles and continued until the discontinuation criteria for treatment were met.

SUMMARY:
This is a Phase 2, multi-center, open-label study to evaluate the efficacy, safety and pharmacokinetics of quizartinib monotherapy in Japanese subjects with FLT3-ITD positive refractory or relapsed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* AML patients in first relapse or refractory after all prior therapy
* Presence of the FLT3-ITD activating mutation in bone marrow or peripheral blood
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* AML secondary to prior chemotherapy for other neoplasms.
* Persistent, clinically significant > Grade 1 non-hematologic toxicity from prior AML therapy
* Prior treatment with a FLT3 targeted therapy
* Active infection not well controlled by antibacterial, antifungal and/or antiviral therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (27):
- Japan (27):
  - Aichi
  - Akita
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Gunma
  - Hiroshima
  - Hokkaido
  - Ibaraki
  - Kagoshima
  - Kanagawa
  - Kyoto
  - Miyagi
  - Nagasaki
  - Nara
  - Okayama
  - Osaka
  - Saga
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokyo
  - Toyama
  - Yamagata
  - Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 participants who met all inclusion and no exclusion criteria were enrolled in the study.
Pre-assignment Details: Quizartinib initial dose was 30 mg/day and escalated to 60 mg/day. For subjects receiving strong cytochrome P450 (CYP) 3A4 inhibitors, the initial dose was 20 mg/day. An increase from the initial dose of 30 mg/day to 60 mg/day or 20 mg/day to 30 mg/day was determined on Day 16 of Cycle 1 and Day 1 of Cycle 2 based on dose increase criteria.
Period: Overall Study
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib
Started | 34 | 3
Completed | 9 | 0
Not Completed | 25 | 3
Not completed — Required stem cell transplant | 13 | 2
Not completed — Progressive disease | 11 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 34 | 3 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 2 | 17
  >=65 years | 19 | 1 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (14.51) | 58.0 (9.92) | 60.0 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 0 | 22
  Male | 12 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 3 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 34 | 3 | 37
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.72 (2.53) | 22.25 (3.37) | 20.84 (2.58)
FLT3-ITD Status [Count of Participants; unit: Participants]
  Positive | 29 | 3 | 32
  Negative | 5 | 0 | 5
Response to Prior Therapy [Count of Participants; unit: Participants]
  Relapse | 21 | 3 | 24
  Refractory | 13 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Composite Complete Remission (CRc) Rate After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: The composite complete remission (CRc) rate is defined as the proportion of participants whose best response is complete remission [CR], CR with incomplete platelet recovery [CRp], or CR with incomplete hematological recovery [CRi]) after treatment with quizartinib.
Time Frame: Baseline, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 up until the end of treatment, except for responses from any subsequent AML therapy including transplantation
Population: All participants with FLT3-ITD positive relapsed or refractory AML who achieved CR, CRp, or CRi, discontinued the study treatment, or completed response assessment at Cycle 4 Day 1.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Total: All participants who received either 30 mg/day or 20 mg/day quizartinib as an initial dose.
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 23 | 3 | 26
percentage of participants | 56.5 [37.5 to 74.2] | 33.3 [1.7 to 86.5] | 53.8 [36.2 to 70.8]

2. Secondary Outcome: Best Response After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: Best response is defined as the best measured response over all response assessments (complete response [CR], CR with incomplete platelet recovery [CRp], CR with incomplete hematological recovery [CRi], partial remission [PR], no response [NR], or Unknown) at all time points after the first dose of the study drug to the end of treatment (does not include response from any subsequent AML therapy including transplantation).
Time Frame: Baseline, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 until the end of treatment, except for responses from any subsequent AML
Population: All participants with FLT3-ITD positive relapsed or refractory AML who achieved CR, CRp, CRi, or PR, discontinued the study treatment, or completed response assessment at Cycle 4 Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 24 | 3 | 27
Participants
  Complete response (CR) | 0 | 0 | 0
  Complete response with incomplete platelet (CRp) | 1 | 0 | 1
  Complete response with incomplete hematologic(CRi) | 12 | 1 | 13
  Partial remission (PR) | 6 | 1 | 7
  No response (NR) | 5 | 1 | 6

3. Secondary Outcome: Response Rate After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 24 | 3 | 27
percentage of participants | 79.2 [57.8 to 92.9] | 66.7 [9.4 to 99.2] | 77.8 [57.7 to 91.4]

4. Secondary Outcome: Duration of Composite Complete Remission (CRc) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: Duration from the date of first composite complete remission (CRc) (complete remission [CR], CR with incomplete platelet recovery [CRp], or CR with incomplete hematological recovery [CRi]) observed to the date of documented relapse was assessed.
Time Frame: as for outcome 1
Population: All participants with FLT3-ITD positive relapsed or refractory AML who had a documented best response of CRc.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 13 | 1 | 14
weeks | 16.1 [4.7 to 24.6] | NA [NA to NA] — A median value was not reached due to <50% of participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | 16.1 [4.7 to 24.6]

5. Secondary Outcome: Overall Survival (OS) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: OS is defined as the time from registration (enrollment) until death from any cause.
Time Frame: Baseline, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 until the end of treatment, except for responses from any subsequent AML therapy including transplantation up to 1 year
Population: All participants with FLT3-ITD positive relapsed or refractory AML.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 29 | 3 | 32
weeks | 34.1 [27.1 to NA] — Upper limit was expressed as NA since the upper limit was not reached. The upper limit was not estimated because of the small number of events after the median OS time. | NA [22.6 to NA] — There were not enough events to estimate a standard error for the median survival time" | 34.1 [27.1 to NA] — Upper limit was expressed as NA since the upper limit was not reached. The upper limit was not estimated because of the small number of events after the median OS time.

6. Secondary Outcome: Event-free Survival (EFS) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: Event-free survival is defined as the time from date of registration until documented refractory disease, relapse after response of composite complete remission (CRc = complete remission [CR], CR with incomplete platelet recovery [CRp], or CR with incomplete hematological recovery [CRi]), or death from any cause, whichever occurs first.
Time Frame: Baseline, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 until the end of treatment, except for responses from any subsequent AML therapy including transplantation up to 32 weeks
Population: All participants with FLT3-ITD positive relapsed or refractory AML.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 29 | 3 | 32
weeks | 12.7 [0.1 to 24.7] | 0.1 [0.1 to NA] — The missing upper bound is related to right-censored data. The last time point censored and estimate is essentially infinity, therefore it is N/A. | 12.7 [0.1 to 24.7]

7. Secondary Outcome: Leukemia-free Survival (LFS) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: Leukemia-free survival (LFS) is the time from the first documented response of CRc until documented relapse or death from any cause. The analysis for LFS will be conditional on the participant having a documented best response of CRc.
Time Frame: Baseline, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 until the end of treatment, except for responses from any subsequent AML therapy including transplantation up to 28 weeks
Population: All participants with FLT3-ITD positive relapsed or refractory AML and documented best response of CRc.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 29 | 3 | 32
weeks | 16.1 [4.7 to 24.6] | NA [NA to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | 16.1 [4.7 to 24.6]

8. Secondary Outcome: Hematopoietic Stem Cell Transplantation Rate After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Description: Proportion of participants who start hematopoietic stem cell transplantation (HSCT) immediately after the end of treatment with the study drug without receiving other treatment for AML, except for conditioning regiment for HSCT, was assessed.
Time Frame: Up to new AML treatment or 1 year post treatment
Population: All participants with FLT3-ITD positive relapsed or refractory AML who underwent HSCT after treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial Dose 20 mg/Day Quizartinib | Total
Number analyzed (Participants) | 29 | 3 | 32
Percentage of participants | 37.9 [20.7 to 57.7] | 33.3 [0.8 to 90.6] | 37.5 [21.1 to 56.3]

9. Secondary Outcome: Change in the Area Under the Plasma Concentration Time Curve (AUC) of Quizartinib and Its Active Metabolite After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Time Frame: Cycle 1, Days 1 and 15; Cycle 2, Day 1
Population: Pharmacokinetic (PK) parameters were assessed in the PK Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Quizartinib 20 mg/Day (With Use of Strong CYP3A4 Inhibitor): Patients who received a CYP3A4 strong inhibitor received quizartinib 20 mg/day and escalated to 30 mg/day at Day 15.
- Quizartinib 30 mg/Day (With No Use of Strong CYP3A4 Inhibitor): Patients who did not receive a CYP3A4 strong inhibitor received quizartinib 30 mg/day.
- Quizartinib 30 mg/Day (With Use of Strong CYP3A4 Inhibitor): Patients who received a CYP3A4 strong inhibitor received quizartinib 30 mg/day.
- Quizartinib 60 mg/Day (With No Use of Strong CYP3A4 Inhibitor): Patients who did not receive a CYP3A4 strong inhibitor received quizartinib 60 mg/day.
Arm/Group | Quizartinib 20 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With No Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 60 mg/Day (With No Use of Strong CYP3A4 Inhibitor)
Number analyzed (Participants) | 3 | 34 | 2 | 21
ng*h/mL
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0): number analyzed (Participants) | 3 | 34 | 0 | 0
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0) | 877 (489) | 1170 (716) |  |
  Cycle 1, Day 1; Active Metabolite (n=3,34,0,0): number analyzed (Participants) | 3 | 34 | 0 | 0
  Cycle 1, Day 1; Active Metabolite (n=3,34,0,0) | 75.1 (80.6) | 560 (391) |  |
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0) | 2610 (693) | 3970 (2610) |  |
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0) | 430 (276) | 3120 (1300) |  |
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21) |  |  | 2960 (749) | 9240 (6090)
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21) |  |  | 983 (389) | 6530 (2630)

10. Secondary Outcome: Change in the Maximum Plasma Concentration (Cmax) of Quizartinib and Its Metabolite (AC886) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Time Frame: Cycle 1, Days 1 and 15; Cycle 2, Day 1
Population: Pharmacokinetic (PK) parameters were assessed in the PK Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quizartinib 20 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With No Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 60 mg/Day (With No Use of Strong CYP3A4 Inhibitor)
Number analyzed (Participants) | 3 | 34 | 2 | 21
ng/mL
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0): number analyzed (Participants) | 3 | 34 | 0 | 0
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0) | 48.1 (25.9) | 76.9 (46.8) |  |
  Cycle 1, Day 1; Active Metabolite (n=3,34,0,0): number analyzed (Participants) | 3 | 34 | 0 | 0
  Cycle 1, Day 1; Active Metabolite (n=3,34,0,0) | 3.92 (4.49) | 29.1 (20.9) |  |
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0) | 127 (35.9) | 211 (132) |  |
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0) | 18.9 (12.1) | 146 (60.4) |  |
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21) |  |  | 149 (38.2) | 480 (296)
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21) |  |  | 43.7 (17.7) | 298 (118)

11. Secondary Outcome: Change in the Trough Plasma Concentration (Ctrough) of Quizartinib and Its Metabolite (AC886) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic (PK) parameters were assessed in the PK Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quizartinib 20 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With No Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 60 mg/Day (With No Use of Strong CYP3A4 Inhibitor)
Number analyzed (Participants) | 3 | 32 | 0 | 0
ng/mL
  Cycle 1, Day 15; Quizartinib | 98.2 (19.7) | 128 (92.5) |  |
  Cycle 1, Day 15; Active Metabolite | 17.8 (11.3) | 112 (47.9) |  |

12. Secondary Outcome: Change in the Time to Reach Maximum Plasma Concentration (Tmax) of Quizartinib and Its Metabolite (AC886) After Treatment With Quizartinib in Japanese Participants With FLT3-ITD Positive Relapsed or Refractory AML
Time Frame: Cycle 1, Days 1 and 15; Cycle 2, Day 1
Population: Pharmacokinetic (PK) parameters were assessed in the PK Analysis Set.
Measure: Median (Full Range); unit: h
Arm/Group | Quizartinib 20 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With No Use of Strong CYP3A4 Inhibitor) | Quizartinib 30 mg/Day (With Use of Strong CYP3A4 Inhibitor) | Quizartinib 60 mg/Day (With No Use of Strong CYP3A4 Inhibitor)
Number analyzed (Participants) | 3 | 34 | 2 | 21
h
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0): number analyzed (Participants) | 3 | 34 | 0 | 0
  Cycle 1, Day 1; Quizartinib (n=3,34,0,0) | 4.08 [2.17 to 6.17] | 4.03 [1.85 to 24.20] |  |
  Cycle 1, Day 1; Active Metabolite (n=2,33,0,0): number analyzed (Participants) | 2 | 33 | 0 | 0
  Cycle 1, Day 1; Active Metabolite (n=2,33,0,0) | 24.33 [24.25 to 24.42] | 24.32 [3.93 to 24.67] |  |
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Quizartinib (n=3,32,0,0) | 4.08 [4.08 to 6.25] | 3.06 [1.42 to 6.08] |  |
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0): number analyzed (Participants) | 3 | 32 | 0 | 0
  Cycle 1, Day 15; Active Metabolite (n=3,32,0,0) | 4.08 [0 to 6.25] | 5.82 [0.83 to 24.50] |  |
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Quizartinib (n=0,0,2,21) |  |  | 6.17 [6.08 to 6.24] | 3.87 [0 to 6.23]
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21): number analyzed (Participants) | 0 | 0 | 2 | 21
  Cycle 2, Day 1; Active Metabolite (n=0,0,2,21) |  |  | 14.17 [4.25 to 24.08] | 5.65 [0 to 24.02]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the informed consent form through 45 days after last dose of study drug up to approximately 2 years.
Description: Adverse events that emerge (or worsen) from the first dose of study drug to the follow-up visit, 45 days after the last dose of study drug, or start date of new AML post treatment.
Groups:
- Initial 20 mg/Day Quizartinib: Participants who received a CYP3A4 strong inhibitor received an initial dose of 20 mg/day of quizartinib and, if no QT prolongation, the dose escalated to 30 mg/day at Day 15.
Arm/Group | Initial Dose 30 mg/Day Quizartinib | Initial 20 mg/Day Quizartinib | Total
All-Cause Mortality (participants affected / at risk) | 13/34 | 1/3 | 14/37
Serious Adverse Events (participants affected / at risk) | 14/34 | 3/3 | 17/37
Other Adverse Events (participants affected / at risk) | 34/34 | 3/3 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose 30 mg/Day Quizartinib (N=34) | Initial 20 mg/Day Quizartinib (N=3) | Total (N=37)
Bacteremia (Infections and infestations) | 2 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hematoma (Vascular disorders) | 1 | 0 | 1
Shock hemorrhagic (Vascular disorders) | 1 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Edema peripheral (General disorders) | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose 30 mg/Day Quizartinib (N=34) | Initial 20 mg/Day Quizartinib (N=3) | Total (N=37)
Acarodermatitis (Infections and infestations) | 3 | 0 | 3
Pneumonia (Infections and infestations) | 3 | 0 | 3
Bacteremia (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 2 | 0 | 2
Device-related infections (Infections and infestations) | 2 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 0 | 10
Anemia (Blood and lymphatic system disorders) | 8 | 1 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Headache (Nervous system disorders) | 4 | 0 | 4
Dysgeusia (Nervous system disorders) | 3 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 3
Hypotension (Vascular disorders) | 1 | 1 | 2
Phlebitis (Vascular disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 9 | 2 | 11
Vomiting (Gastrointestinal disorders) | 6 | 0 | 6
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 4
Constipation (Gastrointestinal disorders) | 2 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 3
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 2
Liver disorder (Hepatobiliary disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Pyrexia (General disorders) | 4 | 1 | 5
Edema (General disorders) | 2 | 1 | 3
Malaise (General disorders) | 2 | 0 | 2
Edema peripheral (General disorders) | 2 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 12 | 1 | 13
Platelet count decreased (Investigations) | 13 | 0 | 13
Neutrophil count decreased (Investigations) | 8 | 0 | 8
White blood cell count decreased (Investigations) | 8 | 0 | 8
Alanine aminotransferase increased (Investigations) | 4 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 3
Liver function test increased (Investigations) | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2
Blood uric acid increased (Investigations) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02984995/Prot_SAP_000.pdf